CLINICAL TRIAL: NCT03005002
Title: A Pilot Feasibility Study of Durvalumab (MEDI4736) and Tremelimumab Following Radioembolization in Patients With Metastatic Microsatellite Stable (MSS) Colorectal Cancer to the Liver
Brief Title: Durvalumab and Tremelimumab in Treating Patients With Microsatellite Stable Metastatic Colorectal Cancer to the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16423; NCI-2016-02001 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16423 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Carcinoma in the Liver; MLH1 Gene Mutation; MSH6 Gene Mutation; PMS2 Gene Mutation; Stage IV Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, tremelimumab) (Experimental): Patients receive durvalumab IV over 60 minutes and tremelimumab IV over 60 minutes on day 1. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Beginning at week 17, patients receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 4 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This pilot clinical trial studies the side effects and how well durvalumab and tremelimumab work in treating patients with microsatellite stable colorectal cancer that has spread to the liver. Monoclonal antibodies, such as durvalumab and tremelimumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the safety of durvalumab and tremelimumab following radioembolization with selective internal radiation (SIR)-Spheres in patients with microsatellite stable (MSS) metastatic colorectal cancer to the liver.

II. Determine the hepatic response rate of SIR-Spheres followed by durvalumab and tremelimumab in patients with MSS metastatic colorectal cancer to the liver.

SECONDARY OBJECTIVES:

I. Estimate the progression free survival (PFS) and overall survival (OS) of the overall treated population.

II. Describe the overall response rate of the treated population. III. Describe the extra-hepatic response in the treated population (abscopal responses).

TERTIARY OBJECTIVES:

I. Describe intra-tumor immune alterations following SIR-Spheres, and following durvalumab plus tremelimumab in comparison to baseline through serial hepatic metastases biopsies.

II. Describe the immune alterations in the blood following SIR-Spheres and following durvalumab plus tremelimumab.

OUTLINE:

Patients receive durvalumab intravenously (IV) over 60 minutes and tremelimumab IV over 60 minutes on day 1. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Beginning at week 17, patients receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 4 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the subject and/or legally authorized representative
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of > 12 weeks
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 75 x 10^9/L (>= 75,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional upper limit of normal given that all patients have liver metastases
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: >= 60 years old and no menses for >= 1 year without an alternative medical cause; AND/OR history of hysterectomy, AND/OR history of bilateral tubal ligation, AND/OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Patients must have received at least one prior line of therapy for the treatment of metastatic disease with a fluoropyrimidine in combination with oxaliplatin and/or irinotecan; patients with prior adjuvant therapy who progressed within 6 months of completion of treatment may be eligible
* Patients must have liver-only metastases or predominant liver metastatic disease
* Patients should have microsatellite stable (MSS) tumor by polymerase chain reaction (PCR) assay or mismatch repair protein proficient (MMRP) tumor by immunohistochemistry as confirmed by the presence of MLH1, MSH2, MSH6, and PMS2; the diagnosis of colorectal cancer should be confirmed by pathology either on the primary tumor or from a prior biopsy of a metastatic disease site
* Patients should have been identified by their respective physicians as candidates for radioembolization and scheduled to undergo such a procedure
* Patients should agree to serial liver metastases biopsy pre-treatment, post-radioembolization, and post-combination immunotherapy
* Patients should have measurable metastatic disease in the liver, defined (for the purpose of this study) as at least 1 measurable lesion more than 2 cm in size and readily accessible to ultrasound (US) or computed tomography (CT)-guided biopsy
* Patients should not be deemed candidate for curative hepatic resection

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) or previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 2 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligns without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
* Receipt of the last dose of chemotherapy or tyrosine kinase inhibitors should be at least 3 weeks prior to durvalumab and tremelimumab dosing; monoclonal antibodies such as bevacizumab, ziv-aflibercept, ramucirumab, cetuximab, and panitumumab should be at least 6 weeks prior to durvalumab and tremelimumab therapy
* Clinical ascites
* Liver involvement by > 50% with metastatic disease determined by the investigator
* Complete portal vein thrombosis on CT scans
* Failure to satisfy minimum criteria of lung shunting (> 20%) or presence of extrahepatic gastrointestinal activity on microaggregated albumin (MAA) scan or angiogram that preclude SIR-Spheres
* Prior external beam radiation to the liver
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2) from previous anti-cancer therapy; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior systemic anti-cancer immunotherapy treatment
* Active or prior documented autoimmune disease within the past 2 years; NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
* Subjects with uncontrolled seizures
* Patients with symptomatic extrahepatic metastases
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* Known allergy or hypersensitivity to investigational product (IP) or any excipient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Hepatic tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 1 year
  Will be summarized using a 90% exact Clopper-Pearson confidence interval
Incidence of adverse events assessed by NCI CTCAE version 4.03 | Up to 1 year
  Toxicities observed will be summarized in terms of type and severity.

SECONDARY OUTCOMES:
Extrahepatic disease response assessed by RECIST 1.1 | Up to 1 year
Hepatic PFS | From study treatment to first progression in the treated liver or death (whichever occurs first), assessed up to 1 year
  This will be reported for the overall population (safety analysis set) and will be described for liver only (time to hepatic progress or death) and for overall disease burden (progression free survival per se). Progression free survival will be estimated using the product-limit (Kaplan-Meier) method, with any loss to follow-up as censoring.
OS | From study treatment to death, assessed up to 1 year
  Overall survival will be estimated using the product-limit (Kaplan-Meier) method, with any loss to follow-up as censoring.
Overall PFS | From study treatment to progressive disease (hepatic and extrahepatic) and death, assessed up to 1 year
  This will be reported for the overall population (safety analysis set) and will be described for liver only (time to hepatic progress or death) and for overall disease burden (progression free survival per se). Progression free survival will be estimated using the product-limit (Kaplan-Meier) method, with any loss to follow-up as censoring.
Overall response rate (both hepatic and extrahepatic disease) assessed by RECIST 1.1 | Up to 1 year

OTHER OUTCOMES:
Tumor immune profiling | Up to 1 year
  Will be summarized using standard statistical summaries.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States